CLINICAL TRIAL: NCT05256017
Title: Safety and Tolerability Study of Acoziborole in g-HAT Seropositive Non-parasitologically Confirmed Subjects: a Multicentre Randomised Double-blind Placebo-controlled Study
Brief Title: Safety and Tolerability Study of Acoziborole in g-HAT Seropositive Subjects
Acronym: OXA004
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNDi-OXA-04-HAT
Record Dates: First submitted 2022-01-17; First posted 2022-02-25 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Trypanosomiasis, African; Trypanosoma Brucei Gambiense; Infection; Sleeping Sickness
Keywords: Human African Trypanosomiasis; Trypanosoma Brucei Gambiense; Sleeping sickness; g-HAT; g-HAT seropositive individuals
MeSH Terms: conditions — Trypanosomiasis, African; Infections

STUDY DESIGN:
Intervention Model Description: Unbalanced, randomized (ratio of 3:1 [acoziborole:placebo]) parallel-arm study. Study treatment (acoziborole or placebo) administered on Day 1. Post-treatment hospitalization of 5 days (up to Day 5). Follow-up visits scheduled at Month 1 and Month 4 (End of Study visit).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acoziborole (Experimental): Single dose administration of acoziborole, 3 tablets of 320 mg
  Interventions: Drug: Acoziborole
- Placebo (Placebo Comparator): Single dose administration of acoziborole matching placebo, 3 tablets of 320 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acoziborole — Single dose administration of acoziborole (3 tablets of 320 mg) on Day 1
  Arms: Acoziborole
Drug: Placebo — Single dose administration of placebo (3 tablets of 320 mg) on Day 1
  Arms: Placebo

SUMMARY:
Human African trypanosomiasis (HAT) or sleeping sickness is a tropical disease which is endemic in sub-Saharan Africa. Most cases of HAT are due to the parasite Trypanosoma brucei gambiense (T.b. gambiense), which is transmitted by the bite of the tsetse fly. HAT can be fatal without diagnosis and treatment. Several treatment options are currently available to treat HAT caused by the T.b. gambiense parasite (g-HAT), but these treatments can be administered only after demonstrating via microscopy the presence of the parasite in a body fluid. However, there are factors such as low parasitaemia and the complexity and low sensitivity of parasitological methods that make such demonstration difficult. It has been demonstrated that a variable proportion (mainly depending on the prevalence) of such g-HAT "sero-suspects" are confirmed cases and, therefore, remain potential reservoirs of the parasite and a source of new infections hindering the efforts to eliminate the disease.

The drug acoziborole was evaluated in a study called "DNDi-OXA-02-HAT". During this study, patients with g-HAT from the DRC and Guinea took a single dose of acoziborole. This study showed that acoziborole has a high efficacy and is safe for treating patients with confirmed g-HAT .

The present study is called "DNDi-OXA-04-HAT". It included seropositive participants from the DRC and Guinea who did not have parasites detected via microscopy in a body fluid. Its objective was to collect data on the safety and tolerability of a single dose of acoziborole compared to a placebo (i.e. a dummy treatment). The results of this study would help decide if acoziborole can be used in the population of g-HAT seropositive individuals and help eliminate the HAT disease.

DETAILED DESCRIPTION:
HAT, or sleeping sickness, is a neglected tropical disease which is endemic in sub Saharan Africa. This vector-borne parasitic disease is transmitted by the bite of the tsetse fly and can be fatal without diagnosis and treatment. The parasites responsible for HAT are the protozoa T.b. gambiense and T.b. rhodesiense. In 2021-2022, HAT due to T.b. gambiense (g-HAT) represented 94% of all HAT cases detected.

Between 2018 and 2022, approximately 1.5 million people lived in areas (mainly rural areas of sub-Saharan Africa) considered to be at moderate to very high risk of HAT and where the disease is still considered as a public health problem. Thanks to efforts from national control programs, supported by the World Health Organization (WHO), non-governmental organizations, bilateral cooperations, the private sector (including pharmaceutical companies) and philanthropic organizations, the number of cases of g-HAT is consistently falling. With respectively 799 and 675 cases of g-HAT reported in 2022 and 2023, the global goal of sustainable disease elimination by 2030, including the interruption of g HAT transmission, is achievable. As the numbers of reported cases diminish, resources for surveillance and specialized screening also taper. This decrease, coupled with the loss of diagnostic skills and disease management expertise, could lead to a weak and less specialized HAT technical environment.

Several therapeutic options are currently available to treat g-HAT at either the hemolymphatic (early) stage or meningoencephalitic (late) stage. In December 2018, fexinidazole was registered for the treatment of g-HAT in DRC. Since then, all other endemic countries authorized the use of fexinidazole for the treatment of g-HAT. Fexinidazole is administered as a 10 day oral treatment to patients with early- or late-stage g-HAT. In patients with very advanced g-HAT, nifurtimox eflornithine combination therapy (NECT) remains the first line treatment, due to the increased risk of relapse in these patients when treated with fexinidazole. Children with g-HAT who have a body weight below 20 kg and/or are under 6 years of age are treated with pentamidine (early stage) or NECT (late stage). Pentamidine and NECT are administered as intravenous (IV) infusions performed daily, over 7 days.

Whilst the delivery of fexinidazole has simplified the management of g-HAT and has facilitated the integration of g-HAT treatment into general health systems, it is expected that the current investment in acoziborole as an oral, single-dose treatment will help boost elimination efforts envisioned for all stages of g-HAT. Indeed, treatment with NECT and fexinidazole are conditioned by the demonstration of the parasite in any body fluid via microscopy. However, factors such as low parasitemia as well as the complexity of parasitological diagnostic methods make this demonstration difficult.

Acoziborole, as a single-dose oral administration, was studied in the open-label pivotal Phase II/III study (DNDi-OXA-02-HAT). The study was conducted in patients with g-HAT (all stages) in the DRC and Guinea. The results of the study showed the high efficacy of acoziborole in any stage of g-HAT, which was comparable to the efficacy of the reference treatment NECT used as a yardstick. Safety data collected during this study did not identify any new safety signals. Based on these data, the benefit-risk balance for treating g-HAT patients (regardless of the disease stage) with acoziborole administered as a single oral dose of 960 mg appeared favorable.

The present study (DNDi-OXA-04-HAT) was conducted in g-HAT seropositive individuals who were unconfirmed parasitologically. It was designed with the objective of assessing the safety and tolerability of a single 960-mg dose of acoziborole compared with placebo during a follow-up period of 4 months.

This study included an exploratory Sub-Study named "TrypSkin" which had the main objective of assessing the presence of extravascular dermal T.b. gambiense in the enrolled population. Participation in this Sub-Study was optional.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form (ICF)
* Male or female
* 15 years of age or older
* Card agglutination test for trypanosomiasis (CATT) test or HAT sero-K-set rapid diagnostic test (RDT) positive
* Parasitology negative (in blood and/or lymph node aspirate [if lymphadenopathy is present])
* Karnofsky performance status above 70
* Able to ingest oral tablets
* Known address and/or contact details provided
* Able to comply with the schedule of follow-up visits and other requirements of the study
* Agreement to be hospitalized upon enrolment for at least 5 days (in order to receive in-ward post-treatment observational follow-up through the first 5 days after treatment)
* Agreement to not take part in any other clinical trials during the participation in this study
* For women of childbearing potential:

  * Agreed to have protected sexual relations to avoid becoming pregnant from enrolment up to 3 months after dosing (contraceptive protection was advised and offered at no cost)
  * Negative urine pregnancy tests (before dosing at site level)

Exclusion Criteria:

* Individuals parasitologically confirmed in blood and/or lymph
* Previously treated for g-HAT
* Severe malnutrition, defined as body mass index (BMI) <16 kg/m^2
* Pregnant or breast-feeding women
* For women of childbearing potential:

  * Urine pregnancy test positive
  * Did not accept contraceptive protection (i.e. condom or sexual abstinence) from enrolment up to 3 months after dosing
* Clinically significant medical condition and/or abnormal laboratory results that could, in the opinion of the Investigator, jeopardize the participant's safety or participation in the study

Additional exclusion criteria for the TrypSkin exploratory sub-study:

* Rejection to participate in the exploratory sub-study in the signed ICF
* Known diabetes mellitus
* Known hemophilia

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Kande Betu Kumeso, Dr., Principal Investigator — Ministry of Public Health, Hygiene and Prevention, Kinshasa
Locations (7):
- Democratic Republic of the Congo (6):
  - General Referral Hospital of Bagata, Bagata, Bandundu
  - Hospital of Dipumba, Mbuji-Mayi, East Kasai
  - General Referral Hospital of Idiofa, Idiofa, Kwilu
  - General Referral Hospital of Masi-Manimba, Masi-Manimba, Kwilu
  - General Referral Hospital of Kwamouth, Kwamouth, Mai Ndombe
  - General Referral Hospital of Bandundu, Bandundu Province
- General Referral Hospital of Dubreka, Dubréka, Guinea

RESULTS

PARTICIPANT FLOW:
Groups:
- Acoziborole: Acoziborole: 3 tablets of 320 mg
- Placebo: Acoziborole matching placebo: 3 tablets of 320 mg
Period: Treatment Period
Arm/Group | Acoziborole | Placebo
Started (Randomized and treated) | 907 | 301
Completed (Completed 5-day hospitalization (Safety set)) | 906 | 300
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Follow-up
Arm/Group | Acoziborole | Placebo
Started | 906 | 300
Completed (End of Study visit (Month 4)) | 898 | 298
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set (based on the actual treatment received, determined by the presence/absence of acoziborole in blood)
Groups:
- Placebo: Placebo: 3 tablets of 320 mg
- Total: Total of all reporting groups
Arm/Group | Acoziborole | Placebo | Total
Number analyzed (Participants) | 906 | 300 | 1206
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (17.35) | 36.4 (16.38) | 37.1 (17.11)
Age, Customized [Count of Participants; unit: Participants]
  Adolescent (15-17 years) | 101 | 28 | 129
  Adult (≥18 years) | 805 | 272 | 1077
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 476 | 158 | 634
  Male | 430 | 142 | 572
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 906 | 300 | 1206
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Guinea | 132 | 44 | 176
  Republic of the Congo | 774 | 256 | 1030

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Any TEAEs
Description: Occurrence and excess rate (95% CI) of any TEAEs.
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: Safety set: participants who received at least 1 tablet of the investigational product (based on the actual treatment received, confirmed by drug concentration data).
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 195 | 69
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -1.5, 95% CI 2-sided [-7.2 to 3.7]

2. Primary Outcome: Occurrence of TEAEs - Malaria
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 34 | 14
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Occurrence and excess rate (95% CI) of any TEAEs (by PT, for PTs reported in ≥1% of participants in either arm) from the investigational product administration (Day 1) to the Month 4 follow-up visit; Test type: Other; Excess rate (ER) = -0.9, 95% CI 2-sided [-4.1 to 1.4] — ER: calculated as "occurrence rate of the TEAE in the acoziborole arm" minus "occurrence rate of the TEAE in the placebo arm". CI: calculated using the Wilson score interval

3. Primary Outcome: Occurrence of TEAEs - Acarodermatitis
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 13 | 3
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = 0.4, 95% CI 2-sided [-1.6 to 1.6] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Occurrence of TEAEs - Abdominal Pain
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 23 | 9
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -0.5, 95% CI 2-sided [-3.2 to 1.4] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Occurrence of TEAEs - Enteritis
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 7 | 4
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -0.6, 95% CI 2-sided [-2.6 to 0.6] — [estimate comment as in outcome 2, analysis 1]

6. Primary Outcome: Occurrence of TEAEs - Nausea
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 7 | 3
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -0.2, 95% CI 2-sided [-2.2 to 0.8] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Occurrence of TEAEs - Gastritis
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 6 | 3
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -0.3, 95% CI 2-sided [-2.3 to 0.7] — [estimate comment as in outcome 2, analysis 1]

8. Primary Outcome: Occurrence of TEAEs - Headache
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 53 | 8
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = 3.2, 95% CI 2-sided [0.3 to 5.3] — [estimate comment as in outcome 2, analysis 1]

9. Primary Outcome: Occurrence of TEAEs - Fatigue
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 14 | 5
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -0.1, 95% CI 2-sided [-2.4 to 1.3] — [estimate comment as in outcome 2, analysis 1]

10. Primary Outcome: Occurrence of TEAEs - Blood Potassium Increased
Description: Occurrence and excess rate (95% CI) of common TEAEs (by PT, for PTs reported in ≥1% of participants in either arm).
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 8 | 6
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -1.1, 95% CI 2-sided [-3.5 to 0.3] — [estimate comment as in outcome 2, analysis 1]

11. Primary Outcome: Occurrence of TEAEs by Period of Occurrence
Description: Occurrence and excess rate (95% CI) of any TEAEs, by period of occurrence.
Time Frame: During hospitalization: from investigational product administration (Day 1) to Day 5 (End of Hospitalization); After hospitalization: from Day 5 (discharge) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
participants
  During hospitalization | 124 | 38
  After hospitalization | 106 | 45
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Occurrence and excess rate (95% CI) of any TEAEs reported during hospitalization; Test type: Other; Excess rate (ER) = 1.0, 95% CI 2-sided [-3.7 to 5.1]
Statistical Analysis 2: Comparison: Acoziborole vs Placebo; Occurrence and excess rate (95% CI) of any TEAEs reported after the hospitalization period; Test type: Other; Excess rate (ER) = -3.3, 95% CI 2-sided [-8.2 to 0.9]

12. Primary Outcome: Occurrence of Serious TEAEs
Description: Occurrence and excess rate (95% CI) of any serious TEAEs.
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 3 | 4
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Test type: Other; Excess rate (ER) = -1.0, 95% CI 2-sided [-3.1 to 0.0]

13. Secondary Outcome: Occurrence of Adverse Events (AEs)
Description: Occurrence of any Adverse Event from Inform Consent signature to 4 month follow-up visit.
  Of note, all AEs reported during this study were TEAEs.
Time Frame: From Inform Consent signature (up to 2 days before treatment) to the Month 4 follow up visit (End of Study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 195 | 69
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Of note, all AEs reported during this study were TEAEs; Test type: Other; Excess rate (ER) = -1.5, 95% CI 2-sided [-7.2 to 3.7]

14. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Alanine Aminotransferase
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
U/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 20.6 (7.90) | 20.6 (9.44)
  Day 5 | 21.9 (9.10) | 24.9 (13.42)
  Month 1: number analyzed (Participants) | 883 | 295
  Month 1 | 19.2 (7.87) | 19.5 (11.70)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 20.8 (8.05) | 20.0 (6.71)

15. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Albumin
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
g/dL
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 3.22 (0.471) | 3.23 (0.433)
  Day 5 | 3.12 (0.434) | 3.13 (0.414)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 3.27 (0.413) | 3.24 (0.391)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 3.22 (0.416) | 3.21 (0.398)

16. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Alkaline Phosphatase
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
U/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 99.8 (46.71) | 101.8 (52.59)
  Day 5 | 91.9 (40.18) | 95.7 (46.43)
  Month 1: number analyzed (Participants) | 884 | 294
  Month 1 | 96.6 (47.88) | 98.3 (53.97)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 98.6 (44.85) | 98.1 (49.90)

17. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Aspartate Aminotransferase
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
U/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 32.8 (10.20) | 32.7 (12.41)
  Day 5 | 33.8 (11.21) | 37.2 (19.04)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 31.0 (9.50) | 32.6 (30.32)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 31.8 (10.95) | 31.1 (8.51)

18. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Calcium
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mmol/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 2.314 (0.1341) | 2.322 (0.1216)
  Day 5 | 2.279 (0.1681) | 2.328 (0.1550)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 2.305 (0.1499) | 2.298 (0.1904)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 2.297 (0.1399) | 2.297 (0.1514)

19. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Chloride
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mmol/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 105.3 (3.05) | 105.3 (2.74)
  Day 5 | 105.2 (3.22) | 105.2 (3.53)
  Month 1: number analyzed (Participants) | 883 | 295
  Month 1 | 105.1 (3.04) | 105.0 (3.23)
  Month 5: number analyzed (Participants) | 898 | 298
  Month 5 | 104.8 (2.89) | 104.8 (3.18)

20. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Creatinine
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mg/dL
  Baseline: number analyzed (Participants) | 906 | 298
  Baseline | 0.84 (0.238) | 0.84 (0.230)
  Day 5 | 0.83 (0.256) | 0.81 (0.233)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 0.82 (0.230) | 0.81 (0.220)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 0.81 (0.227) | 0.80 (0.223)

21. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Glucose
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mg/dL
  Baseline: number analyzed (Participants) | 905 | 299
  Baseline | 88.581 (19.9540) | 87.087 (11.3391)
  Day 5 | 89.801 (14.4784) | 89.410 (9.9699)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 91.715 (16.4756) | 90.207 (10.8139)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 91.226 (24.4440) | 89.225 (10.2205)

22. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Potassium
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mmol/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 4.58 (0.537) | 4.60 (0.572)
  Day 5 | 4.67 (0.607) | 4.59 (0.559)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 4.61 (0.589) | 4.60 (0.636)
  Month 4: number analyzed (Participants) | 897 | 298
  Month 4 | 4.59 (0.540) | 4.61 (0.550)

23. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Sodium
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mmol/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 136.7 (3.39) | 136.7 (3.61)
  Day 5 | 137.2 (3.75) | 137.1 (3.97)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 137.2 (3.41) | 137.1 (3.94)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 137.1 (3.36) | 137.0 (3.38)

24. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Total Bilirubin
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mg/dL
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 0.879 (0.3457) | 0.869 (0.3469)
  Day 5 | 0.739 (0.2957) | 0.809 (0.2506)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 0.818 (0.2641) | 0.884 (0.2591)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 0.887 (0.318) | 0.902 (0.2937)

25. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Bicarbonate
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mmol/L
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 27.5 (2.46) | 27.5 (2.60)
  Day 5 | 28.5 (2.39) | 28.2 (2.40)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 28.0 (2.50) | 27.7 (2.44)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 28.0 (2.48) | 27.9 (2.58)

26. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Total Protein
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
g/dL
  Baseline: number analyzed (Participants) | 906 | 299
  Baseline | 7.63 (0.589) | 7.65 (0.565)
  Day 5 | 7.46 (0.566) | 7.61 (0.584)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 7.55 (0.547) | 7.59 (0.583)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 7.54 (0.573) | 7.57 (0.591)

27. Secondary Outcome: Change From Baseline in Biochemistry Parameter: Blood Urea Nitrogen
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
mg/dL
  Baseline: number analyzed (Participants) | 903 | 299
  Baseline | 7.434 (2.5471) | 7.415 (2.6550)
  Day 5: number analyzed (Participants) | 905 | 299
  Day 5 | 8.402 (2.6432) | 8.358 (2.4459)
  Month 1: number analyzed (Participants) | 883 | 295
  Month 1 | 6.951 (2.2998) | 6.820 (2.5365)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 7.501 (2.3841) | 7.383 (2.2759)

28. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
g/dL
  Baseline | 13.09 (1.706) | 13.10 (1.554)
  Day 5 | 12.57 (1.627) | 12.95 (1.513)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 12.78 (1.550) | 13.00 (1.489)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 13.04 (1.644) | 12.93 (1.646)

29. Secondary Outcome: Change From Baseline in Hematology Parameter: Platelet Count
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
10^9 platelets/L
  Baseline | 229.1 (64.75) | 229.0 (63.04)
  Day 5 | 230.5 (65.20) | 226.5 (65.84)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 227.7 (62.55) | 227.6 (64.01)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 228.4 (60.29) | 229.1 (63.44)

30. Secondary Outcome: Change From Baseline in Hematology Parameter: Leukocytes
Description: Changes from baseline to Day 5, Month 1 and Month 4; presented by treatment arm.
Time Frame: From baseline to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 Leukocytes/L
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
10^9 Leukocytes/L
  Baseline | 5.53 (1.576) | 5.46 (1.539)
  Day 5 | 5.64 (1.563) | 5.60 (1.507)
  Month 1: number analyzed (Participants) | 884 | 295
  Month 1 | 5.51 (1.446) | 5.50 (1.427)
  Month 4: number analyzed (Participants) | 898 | 298
  Month 4 | 5.49 (1.385) | 5.52 (1.426)

31. Secondary Outcome: Change From Baseline in ECG (Electrocardiogram) Parameter: Heart Rate (HR)
Description: Actual values at baseline (Day 1 pre-dose) and Day 5. Change from baseline at Day 5 (Δ). Placebo-corrected change from baseline (ΔΔ), calculated using an analysis of covariance (ANCOVA) model adjusted for sex and age.
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: ECG central tendency set: participants who received at least 1 tablet of the investigational product (based on the actual treatment received, confirmed by drug concentration data) and who had valid ECG evaluations.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
beats/min
  Day 1 (pre-dose) | 66.8 (10.7) | 70.0 (12.1)
  Day 5 | 66.4 (9.9) | 69.1 (12.6)
  Change from baseline at Day 5 (Δ) | -0.4 (8.4) | -0.9 (8.3)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -0.4, 90% CI 2-sided [-2.1 to 1.4]

32. Secondary Outcome: Change From Baseline in ECG Parameter: RR Interval
Description: Actual values at baseline (Day 1 pre-dose) and Day 5. Change from baseline at Day 5 (Δ). Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age.
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose) | 921.6 (143.8) | 882.2 (149.3)
  Day 5 | 923.5 (137.4) | 893.7 (149.4)
  Change from baseline at Day 5 (Δ) | 1.9 (103.5) | 11.5 (94.8)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -0.5, 90% CI 2-sided [-22.0 to 21.1]

33. Secondary Outcome: Change From Baseline in ECG Parameter: PR Interval
Description: as for outcome 32
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose): number analyzed (Participants) | 212 | 68
  Day 1 (pre-dose) | 162.4 (25.2) | 162.2 (20.3)
  Day 5: number analyzed (Participants) | 212 | 68
  Day 5 | 161.4 (23.0) | 161.9 (20.5)
  Change from baseline at Day 5 (Δ): number analyzed (Participants) | 212 | 68
  Change from baseline at Day 5 (Δ) | -1.0 (1.11) | -0.3 (12.8)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -1.1, 90% CI 2-sided [-3.6 to 1.3]

34. Secondary Outcome: Change From Baseline in ECG Parameter: QRS Interval
Description: Actual values at baseline (Day 1 pre-dose) and Day 5. Change from baseline at Day 5 (Δ). Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusting for sex and age.
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose) | 82.2 (8.2) | 82.3 (10.2)
  Day 5 | 81.8 (8.4) | 82.5 (9.0)
  Change from baseline at Day 5 (Δ) | -0.5 (5.4) | 0.3 (4.5)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -0.7, 90% CI 2-sided [-1.9 to 0.4]

35. Secondary Outcome: Change From Baseline in ECG Parameter: QT Interval
Description: as for outcome 32
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose) | 389.5 (27.8) | 383.0 (33.1)
  Day 5 | 377.3 (26.7) | 383.1 (30.8)
  Change from baseline at Day 5 (Δ) | -12.1 (21.4) | 0.1 (20.4)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -10.9, 90% CI 2-sided [-15.3 to -6.6]

36. Secondary Outcome: Change From Baseline in ECG Parameter: QTcF
Description: as for outcome 32
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose) | 401.3 (20.0) | 400.5 (24.0)
  Day 5 | 388.5 (20.5) | 399.0 (21.8)
  Change from baseline at Day 5 (Δ) | -12.8 (13.3) | -1.5 (13.8)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -11.5, 90% CI 2-sided [-14.4 to -8.7]

37. Secondary Outcome: Change From Baseline in ECG Parameter: QTcB
Description: as for outcome 32
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 213 | 68
ms
  Day 1 (pre-dose) | 407.9 (23.0) | 410.1 (25.8)
  Day 5 | 394.6 (23.3) | 407.8 (24.6)
  Change from baseline at Day 5 (Δ) | -13.3 (14.2) | -2.3 (14.8)
Statistical Analysis 1: Comparison: Acoziborole vs Placebo; Placebo-corrected change from baseline (ΔΔ), calculated using an ANCOVA model adjusted for sex and age; Test type: Other; Placebo-corrected change from baseline = -11.7, 90% CI 2-sided [-14.9 to -8.6]

38. Secondary Outcome: Placebo-corrected Baseline-adjusted QTcF (ΔΔQTcF), Computed From a Concentration-response (C-R) Model Between Dry Blood Spot Concentration and Changes From Baseline in QTcF Parameter
Description: Mixed linear model developed based on the model defined by Garnett et al (2017).
  The fixed effect parameters of the pre-specified model were intercept, slope for acoziborole concentrations, influence of baseline (centered on mean), and a treatment specific intercept (0=acoziborole, 1=Placebo). Sex and age were included in the model as fixed covariates.
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: C-R analysis set: participants who received at least 1 tablet of the investigational product (based on the actual treatment received, confirmed by drug concentration data), who had valid ECG evaluations, and at least one change from baseline in ECG matching a PK sample.
Measure: Mean (90% Confidence Interval); unit: ms
Arm/Group | Acoziborole
Number analyzed (Participants) | 192
ms | -12.9 [-14.3 to -11.3]
Statistical Analysis 1: Comparison: Acoziborole; Estimated ΔΔQTcF (in ms) computed from a concentration-response (C-R) model between dry blood spot concentration of acoziborole and changes from baseline in QTcF parameter; Test type: Other; Estimate = -10.7, 90% CI 2-sided [-13.5 to -7.85], Standard Deviation 1.72

39. Secondary Outcome: Incidence of Abnormal Values for PR, QRS, QTcB and QTcF According to Pre-defined Thresholds
Description: Incidence of abnormal values for PR, QRS, QTcB and QTcF at Day 1 and/or Day 5, according to pre-defined thresholds
Time Frame: From baseline (Day 1 pre-dose) to Day 5 (End of Hospitalization)
Population: ECG categorical analyses set: participants who received at least 1 tablet of the investigational product (based on the actual treatment received, confirmed by drug concentration data) and who had valid ECG evaluations at Day 1 or Day 5.
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 215 | 68
Participants
  HR <40 beats/min | 0 | 0
  HR >120 beats/min | 0 | 0
  HR relative change from baseline >25% | 6 | 2
  PR >220 ms | 2 | 1
  PR relative change from baseline >25% | 0 | 0
  QRS >120 ms | 1 | 0
  QRS relative change from baseline >25% | 0 | 0
  QTcF >450 ms and ≤480 ms | 2 | 1
  QTcF >480 ms and ≤500 ms | 0 | 0
  QTcF >500 ms | 0 | 0
  QTcF change from baseline >30 ms and ≤60 ms | 0 | 0
  QTcF change from >60 ms | 0 | 0
  QTcB >450 ms and ≤480 ms | 3 | 1
  QTcB >480 ms and ≤500 ms | 1 | 0
  QTcB >500 ms | 0 | 0
  QTcB change from baseline >30 ms and ≤60 ms | 1 | 1
  QTcB change from >60 ms | 0 | 0

40. Primary Outcome: Occurrence of Severe Treatment-related TEAEs
Description: Occurrence and excess rate (95% CI) of any serious TEAEs.
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 0 | 0

41. Primary Outcome: Occurrence of Any Treatment-related TEAEs
Description: Occurrence of any treatment-related TEAEs by arm
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants | 59 | 17

42. Primary Outcome: Occurrence of Treatment-related TEAEs by PT
Description: Occurrence of any treatment-related TEAEs by PT and by arm
Time Frame: From the investigational product administration (Day 1) to the Month 4 follow-up visit (End of Study).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoziborole | Placebo
Number analyzed (Participants) | 906 | 300
Participants
  SOC: Nervous system disorders | 28 | 5
  Abdominal pain | 14 | 6
  Fatigue | 8 | 5
  Decreased appetite | 6 | 1
  Nausea | 5 | 2
  Dizziness | 5 | 1
  Hot flush | 3 | 0
  Pyrexia | 2 | 0
  Insomia | 2 | 0
  Vomiting | 1 | 1
  Dysgeusia | 1 | 0
  Diarrhoea | 1 | 0
  Enteritis | 1 | 0
  Dyspepsia | 1 | 0
  Gastrointestinal sounds abnormal | 1 | 0
  Asthenia | 1 | 0
  Electrocardiogram QT prolonged | 1 | 0
  Muscle spasms | 1 | 0
  Tachycardia | 0 | 1

ADVERSE EVENTS:
Time Frame: From ICF signature (up to 2 days prior treatment) to Month 4 (end of follow-up)
Description: The primary outcome of this study was the collection of Treatment Emergent Adverse Event (TEAE) (i.e collections of AE from Day 1 (post-treatment) to Month 4 (end of follow-up)) Of note, all AEs reported during this study were TEAEs.
Arm/Group | Acoziborole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/906 | 1/300
Serious Adverse Events (participants affected / at risk) | 3/906 | 4/300
Other Adverse Events (participants affected / at risk) | 137/906 | 45/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acoziborole (N=906) | Placebo (N=300)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acoziborole (N=906) | Placebo (N=300)
Headache (Nervous system disorders) | 53 (54) | 8 (9)
Malaria (Infections and infestations) | 34 (35) | 13 (13)
Abdominal pain (Gastrointestinal disorders) | 23 (23) | 9 (10)
Fatigue (General disorders) | 14 (14) | 5 (5)
Acarodermatitis (Infections and infestations) | 13 (13) | 3 (3)
Blood potassium increased (Investigations) | 8 (8) | 6 (7)
Enteritis (Gastrointestinal disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Gastritis (Gastrointestinal disorders) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
No limitations or caveats were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05256017/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT05256017/SAP_001.pdf